CLINICAL TRIAL: NCT06755905
Title: Application Value of Indocyanine Green Lymphography in Management of Microcystic Lymphatic Malformation of the Tongue
Brief Title: Indocyanine Green Lymphography in Management of Lingual Lymphatic Malformation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Children's Hospital (Other)
Responsible Party: Principal Investigator, Tao Han, Clinical Professor, Nanjing Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NanjingCH0116651
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Lymphatic Malformation
Keywords: indocyanine green; tongue; Lymphatic Malformation
MeSH Terms: conditions — Lymphatic Abnormalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lingual LM with ICGL-guided treatment (Experimental): indocyanine green lymphography guided resection combined with sclerotherapy
  Interventions: Procedure: ICGL-guided treatment
- Conventional treatment (Active Comparator): lingual LM with conventional treatment
  Interventions: Procedure: Conventional Treatment group

INTERVENTIONS:
Procedure: ICGL-guided treatment — Indocyanine green lymphography guided resection combined with sclerotherapy
  Arms: lingual LM with ICGL-guided treatment
Procedure: Conventional Treatment group — Resection with sclerotherapy
  Arms: Conventional treatment

SUMMARY:
To elucidate the application of indocyanine green (ICG) fluorescence angiography in the treatment of childhood tongue cLM (clinically localized malignancy, presumed context here), providing a clearer scientific basis for subsequent targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* No previous intervention
* more than 6 months post-treatment follow-up
* Stage I or Stage IIa

Exclusion Criteria:

* History of iodine allergy
* Syndromic cLM
* Severe liver and kidney dysfunction

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Cured (Reduction in dimension greater than 90%) | From enrollment to the end of treatment at 12 weeks
  Reduction in dimension greater than 90%

CONTACTS AND LOCATIONS:
Locations (1):
- Children's hospital of nanjing medical university, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Han T, Shi L, Huang S, Shen W. Application value of indocyanine green lymphography in the management of stage I/IIA microcystic lymphatic malformation of the tongue. Head Face Med. 2025 Jul 14;21(1):51. doi: 10.1186/s13005-025-00529-2. PMID 40660315